CLINICAL TRIAL: NCT00973869
Title: A Pilot Study of Administration of Curcumin to Determine Colonic Curcumin Tissue Levels in Patients Awaiting Colorectal Endoscopy or Patients With Colorectal Cancer Awaiting Resection
Brief Title: Curcumin in Preventing Colorectal Cancer in Patients Undergoing Colorectal Endoscopy or Colorectal Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000648267; LRI-UL-CURCUMIN; EUDRACT-2007-001971-13; EU-20961
Record Dates: First submitted 2009-09-05; First posted 2009-09-09 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2009-09

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Curcumin; Chromatography, High Pressure Liquid

INTERVENTIONS:
Dietary Supplement: curcumin
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: diagnostic endoscopic procedure
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of curcumin may prevent or treat colorectal cancer.

PURPOSE: This phase I trial is studying the side effects of curcumin in preventing colorectal cancer in patients undergoing colorectal endoscopy or colorectal surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine levels of curcumin and its metabolites in normal colorectal tissue in patients undergoing colorectal endoscopy or colorectal cancer surgery following a 14-day course of curcumin.

Secondary

* To assess the practicality, acceptability, and safety of administering 5 capsules of curcumin daily for 14 days.
* To check the presence of curcumin and its metabolites in peripheral blood and urine.

OUTLINE: Patients receive oral curcumin once daily for 14-28 days. Patients then undergo colorectal endoscopy or resection.

Normal colorectal tissue samples are collected via biopsy for curcumin assay after the last dose of curcumin. Patients also undergo blood and urine sample collection at baseline and after the last dose of curcumin for pharmacokinetic analysis by high performance liquid chromatography.

After completion of study treatment, patients are followed up at 14 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Has a positive fecal occult blood test found during a pilot colorectal cancer screening program
  * Awaiting diagnostic or surveillance colonoscopy
  * Diagnosis of colorectal cancer

PATIENT CHARACTERISTICS:

* Able to return for follow-up tests
* Fertile patients must use effective contraception
* No discrete gastric or duodenal ulcer > 5 mm in the past year

  * Patients with a history of Helicobacter pylori-related peptic ulcer disease are eligible after successfully completing antibiotic treatment for Helicobacter pylori
* No significant medical or psychiatric problem, including significant renal, hepatic, or hematological dysfunction, that would make the patient a poor candidate for this study

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior investigational agents
* No prior pelvic radiotherapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of curcumin in colorectal tissue after treatment

SECONDARY OUTCOMES:
Tolerability and compliance
Presence of curcumin and its metabolites in peripheral blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: William P. Steward, MD, PhD, Principal Investigator — University Hospitals, Leicester
Locations (2):
- United Kingdom (2):
  - St. Mark's Hospital, Harrow, England
  - Leicester Royal Infirmary, Leicester, England